CLINICAL TRIAL: NCT02486796
Title: A Comparison Study to Assess the Value of Naturopathic Medicine Given Immediately and Continuously or Delayed Until Cycle 3 in Combination With Neo-Adjuvant Chemotherapy for Breast Cancer
Brief Title: Immediate or Delayed Naturopathic Medicine in Combination With Neo-Adjuvant Chemotherapy for Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Operational barriers prevent critical specimen analyses from being performed.
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MZ2014018
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Quality of Life
MeSH Terms: interventions — coenzyme Q10; Ubiquinone; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate and Continuous Dosing (Active Comparator): Subjects will be dosed with Reishi mushroom extract, Coenzyme Q10 and Melatonin beginning with Cycle 1 Day 1 of their prescribed neoadjuvant chemotherapy.
  Interventions: Biological: Reishi mushroom extract; Drug: Coenzyme Q10; Drug: Melatonin
- Delayed Dosing (Active Comparator): Subjects will be dosed with Reishi mushroom extract, Coenzyme Q10 and Melatonin beginning with Cycle 3 Day 1 of their prescribed neoadjuvant chemotherapy.
  Interventions: Biological: Reishi mushroom extract; Drug: Coenzyme Q10; Drug: Melatonin

INTERVENTIONS:
Biological: Reishi mushroom extract — Reishi mushroom preparation produced water-ethanol extraction.
  Other Names: Ganoderma lucidum
Drug: Coenzyme Q10 — Preparation of coenzyme Q10
  Other Names: Ubiquinone; Ubidecarenone
Drug: Melatonin — Preparation of melatonin
  Other Names: N-acetyl-5-methoxy tryptamine

SUMMARY:
This study is examine the effect of the addition of naturopathic on immunologic and/or inflammatory parameters and/or quality of life in women receiving neoadjuvant chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Biopsy proven diagnosis of invasive adenocarcinoma of the breast
* Recommendation for neoadjuvant chemotherapy.
* Left Ventricular Ejection Fraction (LVEF) assessment by multigated acquisition scan or echocardiogram within 3 months of entering study
* Blood counts:
* Absolute Neutrophil Count ≥1200 cells/mm^3
* Platelet count ≥100,000/mm^3
* Hemoglobin ≥10g/dL
* Serum creatinine ≤ Upper Limit of Normal (ULN) for the laboratory range
* Total bilirubin ≤ ULN for the laboratory range, unless the patient has an elevation >ULN to 1.5 times the ULN resulting from Gilbert's disease or similar syndrome
* Alkaline phosphatase less than or equal to 2.5 x ULN; and
* Aspartate aminotransferase (AST) less than or equal to 1.5 x ULN for the laboratory range
* If skeletal pain present or alkaline phosphatase >ULN (but less than or equal to 2.5x ULN), bone scan or Positron Emission Tomography (PET) scan must not demonstrate metastatic disease
* AST or alkaline phosphatase greater than ULN, no metastatic disease liver identified by CT, MRI or PET scan
* Able to swallow oral medication
* Willing to forego naturopathic treatment for the first 2 treatment cycles
* Willing to start and continue naturopathic interventions as prescribed
* Willing to forego the use of nutritional or botanical supplements during the study

Exclusion Criteria:

* Stage 4 disease
* Present treatment with Warfarin.
* Synchronous bilateral invasive breast cancer
* Treatment including radiation, chemotherapy, and/or targeted therapy for the currently diagnosed breast cancer prior to entering study
* Any sex hormonal therapy e.g. birth control, ovarian hormone replacement therapy, etc. during participation in the study)
* Continued therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators
* Prior history of breast cancer, including Ductal Carcinoma In Situ (subjects with a history of Lobular Carcinoma In Situ are eligible)
* Prior therapy with chemotherapy or targeted therapy agents for any malignancy
* Cardiac disease that would preclude the use of the certain drugs. This includes but is not confined to:
* Active cardiac disease
* Angina pectoris requiring treatment
* Ventricular arrhythmias except controlled benign premature ventricular contractions
* Conduction abnormality requiring a pacemaker
* Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled by medication
* Clinical significant valvular disease
* History of cardiac disease
* Myocardial infarction
* Congestive heart failure
* Cardiomyopathy
* Uncontrolled hypertension, (blood pressure above 150/90 mm/Hg on antihypertensive treatment)
* History or current symptomatic interstitial pneumonitis or pulmonary fibrosis
* Sensory/motor neuropathy ≥ grade 2
* Malabsorption syndrome, ulcerative colitis, resection the stomach or small bowel, or other disease significantly affecting gastrointestinal function
* Other non-malignant systemic disease precluding treatment with study regimens or required follow up
* Contraindication of corticosteroids
* Administration of an investigational agent within 30 days prior to entering study.
* Administration of therapeutic doses of the supplements being studied including maitake, melatonin and Coenzyme Q10 in the previous 30 days.
* Administration of therapeutic doses of immune modulating botanicals in the previous 30 days.
* Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Shannon, ND, Principal Investigator — Midwestern Regional Medical Center, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing
Started | 3 | 2
Completed | 1 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Quality of Life Score
Description: Subject quality of life as measured by a self-administered questionnaire (0 to 10 Likert scale with 0=No Effect to 10=Worst Effect) at each study visit. The symptoms or impact on activities scored included: Pain, Fatigue, Nausea, Sleep Disturbance, Distress, Shortness of Breath, Memory/Recall Problems, Appetite, Drowsiness, Dry Mouth, Sadness, Vomiting, Numbness, General Activities, Mood, Work, Relationships, Walking or Enjoyment.
Time Frame: Initial visit and study visits at 3-week intervals up to 4 months
Population: One subject in the 'Delayed' arm withdrew consent following Study Visit 2. One subject in the 'Immediate' arm did not complete the Quality of Life Questionnaire at Visit 2. One subject in the 'Delayed' arm did not complete the Quality of Life Questionnaire at Visit 5. One subject in the 'Immediate' Arm withdrew consent prior to completing Visit 5.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing
Number analyzed (Participants) | 3 | 2
units on a scale
  Worst Pain (Visit 1) | 0.7 (0.9) | 2.0 (1.0)
  Worst pain (Visit 2): number analyzed (Participants) | 2 | 2
  Worst pain (Visit 2) | 1.0 (1.0) | 1.0 (0.0)
  Worst Pain (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Pain (Visit 3) | 0.7 (0.9) | 2.0 (0.0)
  Worst Pain (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Pain (Visit 4) | 0.5 (0.5) | 1.0 (0.0)
  Worst Pain (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Pain (Visit 5) | 1.0 (0.0) |
  Worst Fatigue (Visit 1) | 1.0 (0.8) | 1.5 (0.5)
  Worst Fatigue (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Fatigue (Visit 2) | 1.0 (1.0) | 3.5 (1.5)
  Worst Fatigue (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Fatigue (Visit 3) | 1.3 (1.2) | 3.0 (0.0)
  Worst Fatigue (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Fatigue (Visit 4) | 1.5 (0.5) | 1.0 (0.0)
  Worst Fatigue (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Fatigue (Visit 5) | 1.0 (0.0) |
  Worst Nausea (Visit 1) | 0.7 (0.9) | 0.0 (0.0)
  Worst Nausea (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Nausea (Visit 2) | 0.0 (0.0) | 1.0 (0.0)
  Worst Nausea (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Nausea (Visit 3) | 0.3 (0.5) | 1.0 (0.0)
  Worst Nausea (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Nausea (Visit 4) | 0.5 (0.5) | 0.0 (0.0)
  Worst Nausea (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Nausea (Visit 5) | 3.0 (0.0) |
  Worst Sleep Disturbance (Visit 1) | 3.3 (0.9) | 3.0 (1.0)
  Worst Sleep Disturbance (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Sleep Disturbance (Visit 2) | 0.5 (0.5) | 1.0 (1.0)
  Worst Sleep Disturbance (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Sleep Disturbance (Visit 3) | 1.7 (0.5) | 1.0 (0.0)
  Worst Sleep Disturbance (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Sleep Disturbance (Visit 4) | 1.0 (0.0) | 0.0 (0.0)
  Worst Sleep Disturbance (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Sleep Disturbance (Visit 5) | 3.0 (0.0) |
  Worst Sleep Distress (Visit 1) | 2.3 (1.2) | 1.0 (0.0)
  Worst Sleep Distress (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Sleep Distress (Visit 2) | 0.5 (0.5) | 1.0 (1.0)
  Worst Sleep Distress (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Sleep Distress (Visit 3) | 1.0 (0.8) | 0.0 (0.0)
  Worst Sleep Distress (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Sleep Distress (Visit 4) | 0.0 (0.0) | 0.0 (0.0)
  Worst Sleep Distress (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Sleep Distress (Visit 5) | 3.0 (0.0) |
  Worst Shortness of Breath (Visit 1) | 0.0 (0.0) | 0.0 (0.0)
  Worst Shortness of Breath (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Shortness of Breath (Visit 2) | 0.0 (0.0) | 0.0 (0.0)
  Worst Shortness of Breath (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Shortness of Breath (Visit 3) | 0.0 (0.0) | 2.0 (0.0)
  Worst Shortness of Breath (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Shortness of Breath (Visit 4) | 0.0 (0.0) | 0.0 (0.0)
  Worst Shortness of Breath (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Shortness of Breath (Visit 5) | 0.0 (0.0) |
  Worst Memory/Recall (Visit 1) | 0.7 (0.9) | 2.5 (1.5)
  Worst Memory/Recall (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Memory/Recall (Visit 2) | 0.5 (0.5) | 1.0 (0.0)
  Worst Memory/Recall (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Memory/Recall (Visit 3) | 1.0 (0.8) | 2.0 (0.0)
  Worst Memory/Recall (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Memory/Recall (Visit 4) | 0.5 (0.5) | 3.0 (0.0)
  Worst Memory/Recall (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Memory/Recall (Visit 5) | 2.0 (0.0) |
  Worst Appetite (Visit 1) | 0.7 (0.5) | 1.5 (1.5)
  Worst Appetite (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Appetite (Visit 2) | 1.0 (1.0) | 1.5 (1.5)
  Worst Appetite (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Appetite (Visit 3) | 2.0 (2.8) | 0.0 (0.0)
  Worst Appetite (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Appetite (Visit 4) | .05 (.05) | 0.0 (0.0)
  Worst Appetite (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Appetite (Visit 5) | 2.0 (0.0) |
  Worst Drowsiness (Visit 1) | 1.0 (0.8) | 1.5 (0.5)
  Worst Drowsiness (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Drowsiness (Visit 2) | 1.0 (1.0) | 2.5 (1.5)
  Worst Drowsiness (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Drowsiness (Visit 3) | 1.0 (0.8) | 3.0 (0.0)
  Worst Drowsiness (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Drowsiness (Visit 4) | 1.0 (0.0) | 1.0 (0.0)
  Worst Drowsiness (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Drowsiness (Visit 5) | 1.0 (0.0) |
  Worst Dry Mouth (Visit 1) | 0.0 (0.0) | 0.5 (0.5)
  Worst Dry Mouth (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Dry Mouth (Visit 2) | 0.5 (0.5) | 1.5 (1.5)
  Worst Dry Mouth (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Dry Mouth (Visit 3) | 0.7 (0.9) | 0.0 (0.0)
  Worst Dry Mouth (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Dry Mouth (Visit 4) | 0.5 (0.5) | 0.0 (0.0)
  Worst Dry Mouth (Visit 15: number analyzed (Participants) | 1 | 0
  Worst Dry Mouth (Visit 15 | 1.0 (0.0) |
  Worst Sadness (Visit 1) | 1.3 (1.2) | 1.5 (1.5)
  Worst Sadness (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Sadness (Visit 2) | 0.0 (0.0) | 1.5 (1.5)
  Worst Sadness (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Sadness (Visit 3) | 0.3 (0.5) | 0.0 (0.0)
  Worst Sadness (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Sadness (Visit 4) | 0.0 (0.0) | 0.0 (0.0)
  Worst Sadness (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Sadness (Visit 5) | 2.0 (0.0) |
  Worst Vomiting (Visit 1) | 0.0 (0.0) | 0.0 (0.0)
  Worst Vomiting (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Vomiting (Visit 2) | 0.0 (0.0) | 0.0 (0.0)
  Worst Vomiting (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Vomiting (Visit 3) | 0.0 (0.0) | 0.0 (0.0)
  Worst Vomiting (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Vomiting (Visit 4) | 0.0 (0.0) | 0.0 (0.0)
  Worst Vomiting (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Vomiting (Visit 5) | 0.0 (0.0) |
  Worst Numbness (Visit 1) | 0.0 (0.0) | 0.0 (0.0)
  Worst Numbness (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Numbness (Visit 2) | 0.5 (0.5) | 0.0 (0.0)
  Worst Numbness (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Numbness (Visit 3) | 0.7 (0.9) | 0.0 (0.0)
  Worst Numbness (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Numbness (Visit 4) | 1.0 (0.0) | 0.0 (0.0)
  Worst Numbness (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Numbness (Visit 5) | 2.0 (0.0) |
  Worst Effect on General Activities (Visit 1) | 0.0 (0.0) | 2.0 (1.0)
  Worst Effect on General Activities (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Effect on General Activities (Visit 2) | 1.5 (1.5) | 1.0 (0.0)
  Worst Effect on General Activities (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Effect on General Activities (Visit 3) | 1.0 (1.4) | 2.0 (0.0)
  Worst Effect on General Activities (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Effect on General Activities (Visit 4) | 0.5 (0.5) | 0.0 (0.0)
  Worst Effect on General Activities (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Effect on General Activities (Visit 5) | 1.0 (0.0) |
  Worst Mood (Visit 1) | 1.7 (1.7) | 2.0 (2.0)
  Worst Mood (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Mood (Visit 2) | 0.5 (0.5) | 2.0 (1.0)
  Worst Mood (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Mood (Visit 3) | 0.7 (0.5) | 0.0 (0.0)
  Worst Mood (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Mood (Visit 4) | 0.5 (0.5) | 0.0 (0.0)
  Worst Mood (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Mood (Visit 5) | 2.0 (0.0) |
  Worst Effect on Work (Visit 1) | 1.7 (1.2) | 0.0 (0.0)
  Worst Effect on Work (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Effect on Work (Visit 2) | 1.0 (1.0) | 0.5 (0.5)
  Worst Effect on Work (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Effect on Work (Visit 3) | 0.7 (0.9) | 2.0 (0.0)
  Worst Effect on Work (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Effect on Work (Visit 4) | 1.0 (0.0) | 1.0 (0.0)
  Worst Effect on Work (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Effect on Work (Visit 5) | 1.0 (0.0) |
  Worst Effect on Relationships (Visit 1) | 1.0 (1.4) | 0.0 (0.0)
  Worst Effect on Relationships (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Effect on Relationships (Visit 2) | 0.0 (0.0) | 0.0 (0.0)
  Worst Effect on Relationships (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Effect on Relationships (Visit 3) | 0.7 (0.9) | 0.0 (0.0)
  Worst Effect on Relationships (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Effect on Relationships (Visit 4) | 0.5 (0.5) | 0.0 (0.0)
  Worst Effect on Relationships (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Effect on Relationships (Visit 5) | 1.0 (0.0) |
  Worst Walking (Visit 1) | 0.7 (0.9) | 2.0 (2.0)
  Worst Walking (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Walking (Visit 2) | 1.0 (1.0) | 0.5 (0.5)
  Worst Walking (Visit 3): number analyzed (Participants) | 3 | 1
  Worst Walking (Visit 3) | 0.7 (0.7) | 0.0 (0.0)
  Worst Walking (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Walking (Visit 4) | 0.5 (0.5) | 0.0 (0.0)
  Worst Walking (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Walking (Visit 5) | 2.0 (0.0) |
  Worst Effect on Enjoyment (Visit 1) | 0.7 (0.9) | 1.5 (0.5)
  Worst Effect on Enjoyment (Visit 2): number analyzed (Participants) | 2 | 2
  Worst Effect on Enjoyment (Visit 2) | 0.5 (0.5) | 1.0 (0.0)
  1Worst Effect on Enjoyment (Visit 3): number analyzed (Participants) | 3 | 1
  1Worst Effect on Enjoyment (Visit 3) | 0.7 (0.9) | 2.0 (0.0)
  Worst Effect on Enjoyment (Visit 4): number analyzed (Participants) | 2 | 1
  Worst Effect on Enjoyment (Visit 4) | 0.5 (0.5) | 1.0 (0.0)
  Worst Effect on Enjoyment (Visit 5): number analyzed (Participants) | 1 | 0
  Worst Effect on Enjoyment (Visit 5) | 1.0 (0.0) |

2. Secondary Outcome: Concentration of C-reactive Protein in Serum (mg/L)
Description: The serum concentration of C-reactive protein will be measured by approved methods.
Time Frame: Initial visit and study visits at 3-week intervals up to 4 months
Population: C-reactive protein was not determined for one subject in the 'Immediate' Arm at Visit 1, one subject in the 'Delayed' Arm at Visit 2 and one subject in the 'Immediate' Arm at Visit 3 due to blood sample not collected. One subject in each arm withdrew consent after visits 2 and 4, respectively.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing
Number analyzed (Participants) | 3 | 2
mg/dl
  Visit 1: number analyzed (Participants) | 2 | 2
  Visit 1 | 0.20 (0.00) | 0.15 (0.05)
  Visit 2: number analyzed (Participants) | 3 | 1
  Visit 2 | 0.50 (0.12) | 0.03 (0.00)
  Visit 3: number analyzed (Participants) | 2 | 1
  Visit 3 | 0.30 (0.10) | 0.03 (0.00)
  Visit 4: number analyzed (Participants) | 2 | 1
  Visit 4 | 0.40 (0.10) | 0.03 (0.00)
  Visit 5: number analyzed (Participants) | 1 | 1
  Visit 5 | 0.30 (0.00) | 0.10 (0.00)

3. Secondary Outcome: Concentration of Circulating Tumor Cells in Blood (Cells Per Milliliter)
Description: The serum concentration of circulating tumor cells will be measured by approved methods.
Time Frame: Initial visit and study visits at 3-week intervals up to 4 months
Population: Circulating tumor cells were not determined for one subject in the 'Immediate' Arm at Visit 1, one subject in the 'Delayed' Arm at Visit 2 and one subject in the 'Immediate' Arm at Visit 3 due to blood sample not collected. One subject in each arm withdrew consent after visits 2 and 4, respectively.
Measure: Mean (Standard Deviation); unit: cells/ml
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing
Number analyzed (Participants) | 3 | 2
cells/ml
  Visit 1: number analyzed (Participants) | 2 | 2
  Visit 1 | 0.0 (0.0) | 0.0 (0.0)
  Visit 2: number analyzed (Participants) | 3 | 1
  Visit 2 | 0.0 (0.0) | 0.0 (0.0)
  Visit 3: number analyzed (Participants) | 2 | 1
  Visit 3 | 0.0 (0.0) | 0.0 (0.0)
  Visit 4: number analyzed (Participants) | 2 | 1
  Visit 4 | 0.0 (0.0) | 0.0 (0.0)
  Visit 5: number analyzed (Participants) | 1 | 1
  Visit 5 | 0.0 (0.0) | 0.0 (0.0)

4. Secondary Outcome: Sedimentation Rate of Erythrocytes in Blood (mm/hr)
Description: The erythrocyte sedimentation rate will be measured by approved methods.
Time Frame: Initial visit and study visits at 3-week intervals up to 4 months
Population: Sedimentation rate was not determined for one subject in the 'Immediate' Arm at Visit 1, one subject in the 'Delayed' Arm at Visit 2 and one subject in the 'Immediate' Arm at Visit 3 due to blood sample not collected. One subject in each arm withdrew consent after visits 2 and 4, respectively.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing
Number analyzed (Participants) | 3 | 2
mm/hr
  Visit 1: number analyzed (Participants) | 2 | 2
  Visit 1 | 13.5 (9.5) | 17.0 (7.0)
  Visit 2: number analyzed (Participants) | 3 | 1
  Visit 2 | 17.3 (8.3) | 11.0 (0.0)
  Visit 3: number analyzed (Participants) | 2 | 1
  Visit 3 | 20.5 (9.5) | 13.0 (0)
  Visit 4: number analyzed (Participants) | 2 | 1
  Visit 4 | 14.0 (0.0) | 16.0 (0.0)
  Visit 5: number analyzed (Participants) | 1 | 1
  Visit 5 | 13.0 (0.0) | 18.0 (0.0)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event information was solicited from study subjects at each study visit. CTCAE 4.03 was used to grade adverse events.
Arm/Group | Immediate and Continuous Dosing | Delayed Dosing
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT02486796/Prot_SAP_ICF_000.pdf